CLINICAL TRIAL: NCT01876342
Title: Total ExtraPeritoneal (TEP) Versus Open Minimal Suture Repair for Treatment of Sportsman's Hernia/Athletic Pubalgia: A Randomized Multi-center Trial
Brief Title: TEP Versus Open Repair of Sportsman's Hernia
Acronym: sports hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Hannu Paajanen, Professor of Surgery, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27/2013; 27/2013 (Registry Identifier: 27/2013)
Record Dates: First submitted 2013-06-09; First posted 2013-06-12 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Chronic Pain; Bone Marrow Oedema
Keywords: sports hernia; sportsman's hernia; chronic groin pain; open minimal repair; totally extraperitoneal endoscopic technique
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open repair (Experimental): Open minimal repair (OMR) of Sportsman's hernia using 2-0 continuous sutures
  Interventions: Procedure: open repair
- Endoscopic TEP repair (Active Comparator): Totally Endoscopic extraperitoneal repair (TEP)using lightweight mesh
  Interventions: Procedure: endoscopic TEP repair

INTERVENTIONS:
Procedure: open repair — 2-0 sutures
  Arms: Open repair
Procedure: endoscopic TEP repair — mesh
  Arms: Endoscopic TEP repair

SUMMARY:
Sportsman's hernia causes chronic groin pain in physically active adults. Open hernia repair without mesh or laparoscopic technique with mesh have been advocated in the treatment of sportsman's hernia. The aim of this randomized study is to compare the effectiveness of open technique to laparoscopic technique for the treatment of Sportsman´s hernia. The hypothesis is that laparoscopic technique is less painfull than open surgery for repair of sportsman's hernia.

DETAILED DESCRIPTION:
Sportsman's hernia is defined as a weakness or disruption of the posterior wall of the inguinal canal. Open hernia repair with or without mesh or laparoscopic techniques with mesh have been advocated in the treatment of sportsman's hernia and associated athletic pubalgia. The results of the operative treatment from single centers are reported to be good to excellent in between 70 - 90% of patients with the most promising results reported using an open minimal repair (OMR) technique. There are no randomized trials comparing open versus laparoscopic techniques regarding time for recovery and relief of pain. The aim of this randomized study is to compare the effectiveness of OMR technique in local or spinal anesthesia to endoscopic Total ExtraPeritoneal (TEP) technique in general anesthesia for the treatment of Sportsman´s hernia/athletic pubalgia. The primary endpoint is patient being free from intractable groin pain during sports activity or daily work four weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* males/females professional or non-professional athletes
* age 18-50 years
* unilateral or bilateral groin pain lasting > 6 weeks
* physical examination and MRI indicating sportsman's hernia
* pain above inguinal ligament in the deep inguinal ring
* grade I-II edema at pubic symphysis on MRI scan is allowed

Exclusion Criteria:

* patients not willing to participate
* inguinal or femoral hernia
* MRI reveals other major pathology
* former surgery to the actual groin
* allergy to polypropylene or other contra-indication to surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-06; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
pain relief | 4 weeks
  The primary endpoint is number of patients having relief of pain during sports activity (VAS scores 0-20, range 0-100) at four weeks after surgery.

SECONDARY OUTCOMES:
time to training | 3 months
  Secondary end-points are time to resume low-level training and full-level training/competing, complications, one year follow-up and costs of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Paajanen, MD, PhD, Principal Investigator — Kuopio University Hospital, Kuopio, Finland
Locations (1):
- Hannu Paajanen, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Paajanen H, Brinck T, Hermunen H, Airo I. Laparoscopic surgery for chronic groin pain in athletes is more effective than nonoperative treatment: a randomized clinical trial with magnetic resonance imaging of 60 patients with sportsman's hernia (athletic pubalgia). Surgery. 2011 Jul;150(1):99-107. doi: 10.1016/j.surg.2011.02.016. Epub 2011 May 5. PMID 21549403